CLINICAL TRIAL: NCT07051993
Title: A Phase 1, Open-Label, Randomized, Crossover, Two-Part Study to Evaluate the Relative Bioavailability of Two ZN-A-1041 Tablet Formulations Compared to Capsule Formulation and the Effect of Food and Proton Pump Inhibitor on the Pharmacokinetics of ZN-A-1041 Tablet(s) in Healthy Subjects
Brief Title: A Study to Evaluate the Relative Bioavailability of Two Tablet Formulations Compared to Capsule Formulation and the Effect of Food and Proton Pump Inhibitor on ZN-A-1041 Tablet(s) in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: GP45607
Record Dates: First submitted 2025-06-26; First posted 2025-07-04 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Healthy Participants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Part 1: ZN-A-1041 (Experimental): Participants will be administered a single dose of ZN-A-1041 orally.
  Interventions: Drug: ZN-A-1041

INTERVENTIONS:
Drug: ZN-A-1041 — Participants will be administered either a ZN-A-1041 capsule or a tablet orally.

SUMMARY:
This is a Phase 1, open-label, randomized, two-part study to evaluate the relative bioavailability (rBA) of two tablet formulations compared to the capsule formulation of ZN-A-1041 (Part 1). Part 2 of the study will evaluate the effect of food and rabeprazole on the ZN-A-1041 tablet formulation. No participants were enrolled in Part 2 of the study as it has been cancelled.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) within the range of 18 to 32 kg/m^2, inclusive
* Negative hepatitis panel and negative HIV antibody screens
* Negative screening test for latent Mycobacterium tuberculosis infection
* Able to consume the high-fat meal within the protocol-specified time period and willing to consume 100% of the high-fat meal
* Able to fast for 8 hours prior to dosing

Exclusion Criteria:

* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, GI, neurological, or psychiatric disorder
* Personal or family history of congenital long QT syndrome
* History of significant hypersensitivity, intolerance, or allergy to any drug
* History of acute GI symptoms
* History of ophthalmological disease or clinically significant abnormality in the ophthalmic examination
* Have significantly impaired hepatic function
* Female who is pregnant or breastfeeding or intending to become pregnant during the study or within 90 days following the final ZN-A-1041 administration
* Have a QTc interval corrected through use of Fredericia's formula >450 millisecond (msec), PR interval >210 msec, QRS complex >120 msec, or heart rate <50 beats per minute (bpm)
* Use of any drugs known to be moderate or strong inhibitors or inducers of CYP3A or CYP2C8
* Poor peripheral venous access
* History of malignancy within 5 years prior to enrollment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2025-06-27 (Actual); Primary Completion 2025-07-12 (Actual); Study Completion 2025-07-12 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Concentration (Cmax) | Days 1-12 (Part 1)
Area Under the Concentration-Time curve from Hour 0 to the Last Measurable Concentration (AUC0-t) | Days 1-12 (Part 1)
AUC Extrapolated to Infinity (AUC0-inf) | Days 1-12 (Part 1)
Geometric Mean Ratio and Associated 90% Confidence Interval (CI) of Cmax | Days 1-12 (Part 1)
Geometric Mean Ratio and Associated 90% CI of AUC0-t | Days 1-12 (Part 1)
Geometric Mean Ratio and Associated 90% CI of AUC0-inf | Days 1-12 (Part 1)

SECONDARY OUTCOMES:
Time to Maximum Observed Concentration (tmax) | Days 1-12 (Part 1)
Apparent Terminal Elimination Rate Constant | Days 1-12 (Part 1)
Apparent Terminal Elimination Half-Life (t1/2) | Days 1-12 (Part 1)
Apparent Systemic Clearance (CL/F) | Days 1-12 (Part 1)
Apparent Volume of Distribution During the Terminal Elimination Phase (Vz/F) | Days 1-12 (Part 1)
Percentage of Participants With Adverse Events (AEs) | Up to approximately 16 days
Number of Participants With Suicidal Ideation or Suicidal Behavior as Measured Using Columbia-Suicide Severity Rating Scale (C-SSRS) | Baseline, days 1, 5, 9 and 12 (Part 1)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (1):
- Fortrea Leeds CRU, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No